CLINICAL TRIAL: NCT07279779
Title: A Three-Arm Randomized Controlled Trial Evaluating the Efficacy of HypnoDiaCare, an Integrative Hypnosis-Based Diabetes Self-Management Intervention, Compared With EduDiaCare and Neutral Visual Attention Control Among Adults With Type 2 Diabetes Mellitus
Brief Title: HypnoDiaCare Trial: A Randomized Controlled Study of Hypnosis-Integrated Diabetes Self-Management Intervention
Acronym: HDC-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Martaria Rizky Rinaldi, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UGM-PSI-HYPNODIACARE
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Hypnosis; Clinical Hypnosis; Diabetes Self-Management; AADE7 Self-Care Behaviors; Type 2 Diabetes Mellitus; Quality of Life; Randomized Controlled Trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A three-arm, parallel-group randomized controlled trial with pretest-posttest assessments and a delayed-intervention design for the control group.
Who Masked: Participant
Masking Description: Participants were blinded to their group assignment and the specific nature of the intervention they received to minimize expectancy effects. Facilitators could not be blinded due to procedural differences across intervention arms. Outcomes assessors were not involved in intervention delivery and were partially unaware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HypnoDiaCare (Experimental): integrative hypnosis-based diabetes self-management intervention
  Interventions: Behavioral: HypnoDiaCare
- EduDiaCare (Active Comparator): education-only AADE7-based diabetes self-management sessions
  Interventions: Behavioral: EduDiaCare
- Neutral Visual Attention Control (Sham Comparator): neutral visual exposure using standardized non-emotional OASIS images
  Interventions: Other: Neutral Visual Exposure

INTERVENTIONS:
Behavioral: HypnoDiaCare — A two-session individualized behavioral intervention integrating clinical hypnosis with diabetes self-management education. The protocol includes hypnotic induction, deepening, guided imagery, therapeutic suggestion, ego strengthening, and post-hypnotic suggestions, with AADE7 self-care principles embedded within the suggestion phases.
  Arms: HypnoDiaCare
Behavioral: EduDiaCare — A structured two-session diabetes self-management education program based on the AADE7 Self-Care Behaviors framework, covering healthy eating, physical activity, medication adherence, glucose monitoring, emotional coping, decision making, and problem solving. Delivered without hypnosis.
  Arms: EduDiaCare
Other: Neutral Visual Exposure — A two-session presentation of standardized neutral-valence, low-arousal images from the OASIS database. Images are displayed for brief intervals to control for attention and expectancy effects without educational or therapeutic content.
  Arms: Neutral Visual Attention Control

SUMMARY:
This study evaluated the efficacy of HypnoDiaCare, a two-session integrative intervention that combines clinical hypnosis with diabetes self-management education based on the AADE7 Self-Care Behaviors framework, for adults with type 2 diabetes mellitus (T2DM). The trial used a three-arm randomized controlled design with HypnoDiaCare, EduDiaCare (education-only), and a neutral visual attention control group. All participants completed two individual sessions over a 1-2-week interval and completed pretest and posttest assessments.

HypnoDiaCare integrates hypnotic induction, guided imagery, ego strengthening, and positive suggestions with diabetes self-management principles. EduDiaCare provides structured education without hypnosis, and the control group viewed neutral images designed to maintain stable emotional and physiological states.

After the initial posttest, control-group participants were re-randomized to receive HypnoDiaCare or EduDiaCare to explore delayed-intervention effects. Primary outcomes were diabetes self-management and quality of life, while secondary outcomes included psychological symptoms and affective states.

The study aims to determine whether HypnoDiaCare produces greater improvements in self-management and quality of life compared with education-only and attention-control conditions.

DETAILED DESCRIPTION:
This study is a three-arm, pretest-posttest, single-blind randomized controlled trial designed to examine the efficacy of HypnoDiaCare, an integrative intervention combining clinical hypnosis techniques with diabetes self-management education for adults with type 2 diabetes mellitus (T2DM). The trial compared HypnoDiaCare with two comparator conditions: (1) EduDiaCare, a structured education-only program based on the AADE7 Self-Care Behaviors framework, and (2) a neutral visual attention control condition.

Participants were recruited through community health centers (Puskesmas) and social media platforms from December 2024 to March 2025. Eligible participants were adults aged 20 years or older with a documented or self-reported diagnosis of T2DM, able to read Indonesian, and not currently undergoing psychological therapy or experiencing severe psychiatric conditions. All participants provided written informed consent.

Randomization was conducted individually using simple randomization procedures. The study employed a single-blind design in which participants were unaware of the specific nature of the intervention they received. Interventions were delivered individually by trained clinical psychologists following standardized manuals to ensure protocol fidelity.

The HypnoDiaCare intervention consisted of two sessions: a 90-120-minute first session and a 60-minute second session. The structure followed established stages of clinical hypnosis, including induction, deepening, therapeutic imagery, ego strengthening, and post-hypnotic suggestions. Diabetes self-management principles were embedded within the therapeutic suggestion phases. EduDiaCare comprised two 60-minute sessions of individualized diabetes self-management education covering healthy eating, physical activity, medication adherence, glucose monitoring, emotional coping, problem solving, and decision making. The control group received two sessions of neutral visual exposure using standardized affectively neutral images designed to control for attention and expectancy effects.

Primary outcomes were diabetes self-management, assessed using the Indonesian version of the Diabetes Self-Management Instrument (IDN-DSMI), and quality of life measured using the WHOQOL-BREF. Secondary outcomes included depression, anxiety, and stress (DASS-42), as well as affective states measured by the Positive and Negative Affect Schedule - Expanded Form (PANAS-X). Assessments were completed at baseline (pretest) and after the second session (posttest 1). Participants in the control group who later received HypnoDiaCare or EduDiaCare underwent additional pre- and post-intervention assessments for exploratory analysis.

No investigational drugs or devices were used. The study received ethical approval from the Ethics Committee of the Faculty of Psychology, Universitas Gadjah Mada. All procedures were conducted in accordance with ethical standards for research involving human participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 years or older
* Diagnosed with type 2 diabetes mellitus (T2DM), confirmed via self-report or written recommendation from Puskesmas based on medical records
* Able to read and understand Indonesian
* Not currently receiving psychological therapy
* Willing to attend two intervention sessions
* Provided written informed consent

Exclusion Criteria:

* History of severe psychiatric disorders as self-reported
* Currently undergoing psychological treatment or psychotherapy
* Severe physical illness or comorbidities that may interfere with participation
* Cognitive impairment that may hinder comprehension or procedure adherence
* Failure to attend both intervention sessions
* Any condition judged by the investigators to interfere with safe participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Diabetes Self-Management (IDN-DSMI Total Score) | Baseline (pretest) to Posttest 1 (after Session 2), approximately 1-2 weeks
  Diabetes self-management will be assessed using the Indonesian version of the Diabetes Self-Management Instrument (IDN-DSMI), a validated 35-item self-report scale measuring self-integration, self-regulation, interaction with healthcare providers and significant others, glucose monitoring, and treatment adherence. Higher scores indicate better self-management.
Quality of Life (WHOQOL-BREF) | Baseline (pretest) to Posttest 1 (after Session 2), approximately 1-2 weeks
  Quality of life will be measured using the WHOQOL-BREF, a 26-item instrument assessing physical, psychological, social, and environmental domains. Scores are computed using the official WHO scoring method. Higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Depression Symptoms (DASS-42 Depression Subscale) | Baseline to Posttest 1 (~1-2 weeks)
  Assessed using the Depression subscale of the DASS-42, consisting of 14 items rated on a 4-point scale. Higher scores indicate greater depressive symptoms.
Anxiety Symptoms (DASS-42 Anxiety Subscale) | Baseline to Posttest 1 (~1-2 weeks)
  Assessed using the Anxiety subscale of the DASS-42. Higher scores indicate greater anxiety symptoms.
Stress Symptoms (DASS-42 Stress Subscale) | Baseline to Posttest 1 (~1-2 weeks)
  Measured using the General Positive Affect (GPA) composite from the PANAS-X. Higher scores reflect higher positive affect.
Negative Affect (PANAS-X General Negative Affect Score) | Baseline to Posttest 1 (~1-2 weeks)
  Measured using the General Negative Affect (GNA) composite from the PANAS-X. Higher scores reflect higher negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Kwartarini Wahyu Yuniarti, Professor / Ph.D, Study Chair — Gadjah Mada University
Locations (1):
- Hypnotic Guided Imagery Laboratory, Faculty of Psychology, Universitas Gadjah Mada, Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
The plan for sharing individual participant data (IPD) has not yet been finalized. De-identified data may be shared upon reasonable request after primary analyses and publications are completed, subject to ethics approval and data-sharing agreements. No IPD will be shared at this time.